CLINICAL TRIAL: NCT00876967
Title: Comparison of Performance of Three Laryngoscope Blades: Plastic Single Use, Metallic Single Use and Metallic Reusable Blades.
Brief Title: Comparison of Three Laryngoscope Blades for Orotracheal Intubation in the Operating Room
Acronym: Laryngotest
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Hanouz JL PHD, University Hospital, Caen
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Laryngotest; N°ID RCB 2007-A00321-52
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Intubation
Keywords: anesthesiology; randomized; laryngoscope; intubation; laryngeal exposition; laryngoscope blades; plastic single use blade; metallic single use blade; metallic reusable blade; success to intubation at first attempt; Cormack and lehanne modify grade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): metallic single use blade
  Interventions: Device: metallic single use blade
- 2 (Experimental): plastic single use blade
  Interventions: Device: plastic single use blade
- 3 (Active Comparator): metallic reusable blade
  Interventions: Device: metallic reusable blade

INTERVENTIONS:
Device: metallic single use blade — metallic single use blade
  Arms: 1
Device: plastic single use blade — plastic single use blade
  Arms: 2
Device: metallic reusable blade — metallic reusable blade
  Arms: 3

SUMMARY:
The purpose of this study is to determinate if there is a difference in performance provided by three laryngoscope blades: plastic single use, metallic single use and metallic reusable blades.

DETAILED DESCRIPTION:
Primary outcome: success of intubation at the first attempt

Secondary outcomes: quality of laryngeal exposition (Cormack and Lehanne modify grade), duration to success intubation, Intubation difficult Scale and result of intubation procedure

ELIGIBILITY:
Inclusion Criteria:

* patient age over 18 who need general anesthesia with orothracheal intubation

Exclusion Criteria:

* patient age under 18 or major assist
* presence of upper airway malformation or abnormality
* cervical or facial trauma
* previous difficult intubation known
* no use of curare
* Body Mass Index over 30kg/m2 if crush induction use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
success of intubation at the first attempt | immediately

SECONDARY OUTCOMES:
quality of laryngeal exposition (Cormack and Lehanne modify grade) | immediately
duration to success intubation | immediately
Intubation difficult Scale | Immediately
result of intubation procedure | immediately

CONTACTS AND LOCATIONS:
Overall Officials: HANOUZ Jean-Luc, PHD, Study Director — Anesthesiology critical care SAMU departement, University Hospital of Caen
Locations (1):
- University Hospital Caen, Caen, Basse-Normandie, France

REFERENCES:
- [Derived] Buleon C, Parienti JJ, Lesage A, Grandin W, Pouliquen E, Flais F, Simonet T, Gerard JL, Hanouz JL. Comparison of plastic and metallic single-use and metallic reusable laryngoscope blades: a randomised controlled trial. Eur J Anaesthesiol. 2013 Apr;30(4):163-9. doi: 10.1097/EJA.0b013e32835c1cdb. PMID 23274619